CLINICAL TRIAL: NCT06600503
Title: The Effectiveness of a Mobile Lung Rehabilitation System on Patient Satisfaction and Lung Function After Lung Cancer Surgery
Brief Title: The Effect of a Mobile Application on Enhancing Pulmonary Rehabilitation After Lung Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kun-Ling Tsai, Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A-ER-111-055
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Rehabilitation; Telerehabilitation; Lung Cancer
Keywords: pulmonary rehabilitation; mobile application; Telerehabilitation; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- application inttervention group (Experimental): The experimental group will receive standard postoperative care, including chest rehabilitation, a mobile application for remote self-training every day after surgery, and an interactive healthcare web platform for health education.
  Interventions: Behavioral: RehabLung mobile application; Other: Healthcare interactive Web Platform
- Usual care group (Active Comparator): The usual care group will receive standard postoperative care, including chest rehabilitation and an interactive healthcare web platform for health education
  Interventions: Behavioral: Lung cancer postoperative standard care; Other: Healthcare interactive Web Platform

INTERVENTIONS:
Behavioral: RehabLung mobile application — Participants in the intervention group will receive in-person pulmonary rehabilitation during their surgical admission and access to a mobile pulmonary rehabilitation application for self-training. This program begins one month before surgery and continues for seven weeks after surgery. The application is designed to encourage participants to engage in pulmonary rehabilitation exercises from preoperative preparation through postoperative care. It offers guided chest breathing exercises, using visual and movement instructions created and remotely prescribed by a physical therapist. Participants will receive daily breathing exercise prescriptions throughout the study period.
  Other Names: The application group; RehabLung App
  Arms: application inttervention group
Behavioral: Lung cancer postoperative standard care — Participants in the usual care group will receive in-person pulmonary rehabilitation during surgical admission, pre-operative healthcare, and guidance on breathing exercises to practice before surgery. They will also receive post-operative breathing exercise prescriptions to follow at home.
  Other Names: usual care; Standard chest rehabilitation
  Arms: Usual care group
Other: Healthcare interactive Web Platform — The healthcare interactive Web Platform provides patients with surgical information through animations. This includes an introduction to lung surgery, preparation procedures, answers to common patient questions, post-surgery wound care, and a brief guide to pulmonary rehabilitation.

SUMMARY:
The goal of this clinical trial is to investigate the effect of a mobile application intervention on postoperative lung rehabilitation. The main purposes of this study are:

1. To understand the effectiveness of the pulmonary rehabilitation mobile application in improving lung function.
2. To assess the feasibility of the pulmonary rehabilitation mobile application in post-surgery rehabilitation care.

Researchers will compare the intervention group (using the pulmonary rehabilitation mobile application) to the usual care group to determine if the mobile application is effective in lung surgery rehabilitation.

Participants will join the study immediately after providing informed consent and will continue for up to 7 weeks post-surgery. Participants will be randomly allocated to either the intervention group or the control group. Both groups will receive regular pulmonary rehabilitation during their hospital stay (1 day before surgery and 2 to 3 days after surgery). Researchers will guide participants in the intervention group to use the mobile application for pulmonary rehabilitation exercises throughout the study period. Participants in the usual care group will receive health education and an exercise guide before discharge. Participants will undergo three study assessments: at baseline (within 1 week after enrollment), post-surgery (week 5), and at follow-up (week 8).

ELIGIBILITY:
Inclusion Criteria:

* age over 20 years
* primary diagnosis of lung cancer at any stage and type
* referral to lung cancer resection by thoracotomy or videothoracoscopy
* ability to understand and consent to the trial procedures
* conscious and cognition intact

Exclusion Criteria:

* included adjuvant treatments (chemotherapy or radiotherapy)
* previous history of thoracic surgery
* neurological and/or musculoskeletal comorbidities
* visual or hearing impairment
* acute respiratory illness

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity-oxygen consumption | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Cardiorespiratory fitness is evaluated by a cardiopulmonary exercise test using a cycle ergometer. Participants will be encouraged to perform a cycle ergometer stress test to assess their cardiopulmonary function. During the test, the workload will gradually increase by 10 watts per minute until the participant reaches peak exercise capacity. Throughout the exercise test, participants will be carefully monitored for echocardiography and heart rate, and will wear a mask to analyze ventilatory outcomes using a computed gas analysis system. Peak oxygen consumption (VO2 peak) will be measured during the exercise test, and values for the difference and change in percent predicted (peak oxygen uptake [mL/kg/min], VO2 peak difference [mL/kg/min], VO2 peak change [%], and [% predicted]) will be obtained from gas analysis. The predicted values will be referenced from the system based on race, age, height, biological sex, and weight.
Exercise capacity-workload | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Cardiorespiratory fitness is evaluated by a cardiopulmonary exercise test using a cycle ergometer. Participants will be encouraged to perform a cycle ergometer stress test to assess their cardiopulmonary function. During the test, the workload will gradually increase by 10 watts per minute until the participant reaches peak exercise capacity. Throughout the exercise test, participants will be carefully monitored for echocardiography and heart rate, and will wear a mask to analyze ventilatory outcomes using a computed gas analysis system.
  The workload achieved during exercise test will be recored by peak work rate (watts), and peak work rate (%pred.) The predicted workload will be referenced from the system based on race, age, height, biological sex, and weight.
Exercise capacity-ventilatory efficiency | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Cardiorespiratory fitness is evaluated by a cardiopulmonary exercise test using a cycle ergometer. Participants will be encouraged to perform a cycle ergometer stress test to assess their cardiopulmonary function. During the test, the workload will gradually increase by 10 watts per minute until the participant reaches peak exercise capacity. Throughout the exercise test, participants will be carefully monitored for echocardiography and heart rate, and will wear a mask to analyze ventilatory outcomes using a computed gas analysis system.
  The gas analysis of oxygen exchange efficiency includes maximal ventilation (L/min), maximal ventilation (% predicted), ventilatory equivalents slope, VE/VCO2 slope, ventilatory equivalents, and VE/VCO2 (% predicted).
Exercise capacity-Anaerobic threshold | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Cardiorespiratory fitness is evaluated by a cardiopulmonary exercise test using a cycle ergometer. Participants will be encouraged to perform a cycle ergometer stress test to assess their cardiopulmonary function. During the test, the workload will gradually increase by 10 watts per minute until the participant reaches peak exercise capacity. Throughout the exercise test, participants will be carefully monitored for echocardiography and heart rate, and will wear a mask to analyze ventilatory outcomes using a computed gas analysis system.
  Anaerobic threshold (AT) (mL/kg/min) is defined as a nonlinear increase in CO2 production, which will be analyze during gas analysis in an incremental exercise test.
Pulmoanry function | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  The pulmonary function test, assessed by spirometry, is performed to evaluate lung volumes over time and ventilatory capacity. Participants will be guided by experienced therapists to take a maximal inspiration, then exhale with maximal effort for as long and as fast as possible. Measurements include forced vital capacity (FVC [L, % predicted]), forced expiratory volume in one second (FEV1 [L, % predicted]), and the ratio of the two volumes (FEV1/FVC [% predicted]). The predicted values will be referenced from large population studies of healthy adults, matched by race, age, height, biological sex, and weight.

SECONDARY OUTCOMES:
Global respiratory muscle strength | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Global respiratory muscle strength is assessed using a pressure gauge and a mouthpiece. Participants are guided to perform maximal exhalation followed by full inhalation, and then maximal inhalation followed by full exhalation through the mouth. Measurements include maximal inspiratory pressure (PImax [cmH2O, % predicted]) and maximal expiratory pressure (PEmax [cmH2O, % predicted]).
Six Minute Walk Test, 6MWT | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  The six-minute walk test is conducted by having a therapist encourage the participant to walk continuously at a comfortable speed for six minutes. The distance covered during the six-minute walk test (m) will be recorded. Throughout the test, vital signs will be carefully monitored.
Postoperative pulmonary complications | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Postoperative pulmonary complications (PPCs) will be recorded from medical records including atelectasis, pneumothorax, respiratory infection, respiratory failure, pleural effusion, bronchospasm, aspiration pneumonitis, acute respiratory distress syndrome,
Quality of life - EORTC QLQ-C30 | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Quality of life specific to lung cancer patients is assessed using the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30). This questionnaire evaluates various aspects of quality of life, including physical, role, cognitive, emotional, and social functioning, as well as cancer-related symptoms and overall health status. Scores range from 0 to 100 across the 30 items. A higher score on the global scale indicates a better quality of life.
Qulaity of life-WHOQOL-BREF | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  The measurement of quality of life in participants is assessed using the WHOQOL-BREF questionnaire (World Health Organization Quality of Life Brief Version). This questionnaire includes 26 items that assess perceptions of quality of life across physical, psychological, social, and environmental domains, with scores ranging from 0 to 100. Higher scores indicate better quality of life.

OTHER OUTCOMES:
Demographic data | Baseline, post-surgery assessment at week 5, follow-up assessment at week 8
  Body mass index (Kg/m2) Age (years) Sex Smoking (%) (current smokers, never smoked, past smokers) Smoking history (packs/year) Presence of COPD Surgery (lobectomy, minor resection, pneumonectomy) Surgery type (thoracotomy, videothoracoscopy) Histological feature (adenocarcinoma, squamous cell carcinoma, other) Length of hospitalization
Adherence | Post-surgery assessment will be conducted at week 5, followed by a follow-up assessment at week 8.
  Compliance will be assessed using a self-reported questionnaire that tracks participants' adherence to the protocol instructions related to breathing exercises, including frequency, technique, duration, and consistency. This self-reported questionnaire includes 28 scaled questions using a 5-point Likert scale, along with one open-ended question to capture any barriers to compliance or reasons for not following the protocol. The compliance score will be calculated based on participants' responses to the scaled questions and will be expressed as a total compliance score, with higher scores indicating better compliance. The measurement tool will be a customized compliance scale designed for this study, allowing participants to indicate the extent to which they followed the exercise instructions as prescribed.
Compliance | Post-surgery assessment will be conducted at week 5, followed by a follow-up assessment at week 8.
  Compliance will be assessed using a self-reported questionnaire that tracks participants' adherence to the protocol instructions related to breathing exercises, including frequency, technique, duration, and consistency. This self-reported questionnaire includes 28 scaled questions using a 5-point Likert scale, along with one open-ended question to capture any barriers to compliance or reasons for not following the protocol. The compliance score will be calculated based on participants' responses to the scaled questions and will be expressed as a total compliance score, with higher scores indicating better compliance. The measurement tool will be a customized compliance scale designed for this study, allowing participants to indicate the extent to which they followed the exercise instructions as prescribed

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be decided after summarized data being published.